CLINICAL TRIAL: NCT02186509
Title: Phase I Study of Alisertib With Concurrent Fractionated Stereotactic Radiation Treatment for Recurrent High Grade Gliomas
Brief Title: Alisertib and Fractionated Stereotactic Radiosurgery in Treating Patients With Recurrent High Grade Gliomas
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sidney Kimmel Cancer Center at Thomas Jefferson University (Other)
Collaborators: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Thomas Jefferson University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13P.528; 2013-12 (Other: CCRRC); JT 3007 (Other: JeffTrial Number)
Record Dates: First submitted 2014-07-07; First posted 2014-07-10 (Estimated); Results first posted 2019-09-09 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Adult Anaplastic Astrocytoma; Adult Anaplastic Ependymoma; Adult Anaplastic Oligodendroglioma; Adult Brain Stem Glioma; Adult Diffuse Astrocytoma; Adult Giant Cell Glioblastoma; Adult Glioblastoma; Adult Gliosarcoma; Adult Mixed Glioma; Adult Oligodendroglioma; Adult Pilocytic Astrocytoma; Adult Pineal Gland Astrocytoma; Adult Subependymal Giant Cell Astrocytoma; Recurrent Adult Brain Tumor
MeSH Terms: conditions — Astrocytoma; Ependymoma; Oligodendroglioma; Glioblastoma; Gliosarcoma; Glioma; Brain Neoplasms | interventions — Radiosurgery; MLN 8237

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Alisertib, fractionated stereotactic radiosurgery (Experimental): CONCURRENT PHASE: Patients undergo fractionated stereotactic radiosurgery QD every weekday for 10 days and receive alisertib PO BID concurrently with radiation therapy for 10 days.
  MAINTENANCE PHASE: Patients receive alisertib PO BID on days 1-7. Treatment repeats every 21 days for up to 18 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Radiation: Hyperfractionated radiation therapy; Radiation: Stereotactic radiosurgery; Drug: Alisertib; Procedure: Quality-of-life assessment

INTERVENTIONS:
Radiation: Hyperfractionated radiation therapy — Undergo hyperfractionated radiation therapy
Radiation: Stereotactic radiosurgery — Undergo stereotactic radiosurgery
Drug: Alisertib — Given PO
  Other Names: MLN8237
Procedure: Quality-of-life assessment — Ancillary studies

SUMMARY:
This phase I trial studies the side effects and best dose of alisertib when combined with fractionated stereotactic radiosurgery in treating patients with high-grade gliomas that have returned after previous treatment with radiation therapy (recurrent). Alisertib may stop the growth of tumor cells by blocking an enzyme needed for the cells to divide. Radiation therapy uses high energy x rays to kill tumor cells. Stereotactic radiosurgery uses special positioning equipment to send a single high dose of radiation directly to the tumor and cause less damage to normal tissue. Delivering stereotactic radiosurgery over multiple doses (fractionation) may cause more damage to tumor tissue than normal tissue while maintaining the advantage of its accuracy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Evaluate the safety and tolerability of the study treatment. II. To determine the maximum tolerated dose (MTD) of daily oral alisertib when combined with fractionated stereotactic radiation treatment for recurrent high grade glioma.

SECONDARY OBJECTIVES:

I. To estimate 6 month progression free survival rate. II. To estimate the median time to progression. III. To estimate overall survival. IV. To estimate the impact on quality of life (QoL).

OUTLINE: This is a dose-escalation study of alisertib.

CONCURRENT PHASE: Patients undergo fractionated stereotactic radiosurgery once daily (QD) every weekday for 10 days and receive alisertib orally (PO) twice daily (BID) concurrently with radiation therapy for 10 days.

MAINTENANCE PHASE: Patients receive alisertib PO BID on days 1-7. Treatment repeats every 21 days for up to 18 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 1 year and then every 4-6 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have a previously histologically or cytologically confirmed high grade glioma (astrocytic or oligodendroglial supratentorial tumors grade 3 or 4) that has been previously treated with fractionated radiation therapy and now shows evidence of recurrence.
2. Patients must have recovered from the toxic effects of prior therapy.
3. Patients must have recovered from the effects of surgery. There must be a minimum of 21 days from the day of surgery to the day of protocol treatment. For core or needle biopsy, a minimum of 7 days must have elapsed prior to the day of protocol treatment.
4. Prior treatment with cytotoxic and biological agents is permissible. There should be at least a 2-week break between prior treatment and the protocol treatment.
5. Prior treatment with fractionated radiation therapy (up to 60Gy) is an eligibility criterion, however there should not have been a second course of fractionated radiotherapy to the supratentorial area.
6. One prior single fraction radiosurgical procedure within the treatment field is acceptable if V12<5 cc (V12 is the volume of normal brain (outside GTV) receiving 12 or more Gy). Additional radiosurgical procedures outside of the treatment area are acceptable.
7. Subject must be able to take oral medication and to maintain a fast, is required for 2 hours before and 1 hour after MLN8237 administration.
8. ANC > 1500/mm³, platelets > 100,000/mm³, Hgb > 9 g/dL. Values must be obtained without need for myeloid growth factor or platelet transfusion support within 14 days of registration. However, erythrocyte growth factor is allowed as per published ASCO guidelines.
9. Total bilirubin ≤ ULN, SGOT (AST) and SGPT (ALT)< 1.5 x ULN, within 14 days of registration.
10. Adequate renal function as defined by: calculated creatinine clearance must be ≥40 mL/minute (Cockcroft-Gault), within 14 days of registration.
11. Age >18 years.
12. ECOG performance status <2 (see Appendix I).
13. Life expectancy of greater than 2 months.
14. Women of childbearing potential must have a negative β-HCG pregnancy test documented within 7 days prior to registration.
15. Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for 4 months after last dose.
16. Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

1. Known history of uncontrolled sleep apnea syndrome and other conditions that could result in excessive daytime sleepiness such as severe chronic obstructive pulmonary disease requiring supplemental oxygen.
2. Systemic infection requiring IV antibiotic therapy within 14 days preceding the first dose of study drug, or other severe infection.
3. Myocardial infarction within 6 months prior to enrollment, New York Heart Association (NYHA) Class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities. Prior to study entry, any ECG abnormality at Screening has to be documented by the investigator as not medically relevant.
4. Female subject is pregnant or breast-feeding. Confirmation that the subject is not pregnant must be established by a negative serum β-human chorionic gonadotropin (β-hCG) pregnancy test result obtained during screening. Pregnancy testing is not required for post-menopausal or surgically sterilized women.
5. Patient has received other investigational drugs within 14 days before enrollment
6. Serious medical or psychiatric illness likely to interfere with participation in this clinical study.
7. Other severe acute or chronic medical or psychiatric condition, including uncontrolled diabetes, malabsorption, resection of the pancreas or upper small bowel, requirement for pancreatic enzymes, any condition that would modify small bowel absorption of oral medications, or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for enrollment in this study.
8. Treatment with clinically significant enzyme inducers, such as the enzyme-inducing antiepileptic drugs phenytoin, carbamazepine or phenobarbital, or rifampin, rifabutin, rifapentine or St. John's wort within 14 days prior to the first dose of MLN8237 and during the study.
9. Known history of human immunodeficiency virus (HIV) infection, hepatitis B, or hepatitis C. Testing is not required in the absence of clinical findings or suspicion.
10. Patients have a history of any other malignancy from which the patient has been disease-free for less than 2 years, with the exception of adequately treated basal or squamous cell carcinoma of skin, superficial bladder cancer or carcinoma in situ of cervix, AJCC (version 7.0) stage 0 or I breast cancer, AJCC (version 7.0) stage I, or II prostate cancer.
11. Radiation therapy to more than 25% of the bone marrow. Whole pelvic radiation is considered to be over 25%.
12. Patients who cannot swallow whole tablets (i.e. medication tablets)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2015-01-30 (Actual); Primary Completion 2017-03-31 (Actual); Study Completion 2018-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wenyin Shi, MD, PhD, Principal Investigator — Thomas Jefferson University
Locations (1):
- Sidney Kimmel Cancer Center at Thomas Jefferson University, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Song A, Andrews DW, Werner-Wasik M, Kim L, Glass J, Bar-Ad V, Evans JJ, Farrell CJ, Judy KD, Daskalakis C, Zhan T, Shi W. Phase I trial of alisertib with concurrent fractionated stereotactic re-irradiation for recurrent high grade gliomas. Radiother Oncol. 2019 Mar;132:135-141. doi: 10.1016/j.radonc.2018.12.019. Epub 2019 Jan 4. PMID 30825962
- See also: Kimmel Cancer Center at Thomas Jefferson University, an NCI-Designated Cancer Center — https://www.jeffersonhealth.org/clinical-specialties/cancer
- See also: Thomas Jefferson University Hospitals — http://www.JeffersonHospital.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Alisertib, Fractionated Stereotactic Radiosurgery: CONCURRENT PHASE: Patients undergo fractionated stereotactic radiosurgery QD every weekday for 10 days and receive alisertib PO BID concurrently with radiation therapy for 10 days.
  MAINTENANCE PHASE: Patients receive alisertib PO BID on days 1-7. Treatment repeats every 21 days for up to 18 courses in the absence of disease progression or unacceptable toxicity.
  Hyperfractionated radiation therapy: Undergo hyperfractionated radiation therapy
  Stereotactic radiosurgery: Undergo stereotactic radiosurgery
  Alisertib: Given PO
  Quality-of-life assessment: Ancillary studies
Period: Overall Study
Arm/Group | Alisertib, Fractionated Stereotactic Radiosurgery
Started | 17
Completed | 17
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Alisertib, Fractionated Stereotactic Radiosurgery
Number analyzed (Participants) | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 15
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 17
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 17

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) of Alisertib
Description: Defined as the dose at which >= 2 patients experience dose-limiting toxicity, graded in severity according to the National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0
Time Frame: Up to 30 days after completion of radiation therapy
Measure: Number; unit: mg dose of Alisertib
Arm/Group | Alisertib, Fractionated Stereotactic Radiosurgery
Number analyzed (Participants) | 17
mg dose of Alisertib | 50

2. Secondary Outcome: Number of Participants With Complete or Partial Response
Description: 95% confidence intervals will be computed. Response was defined by the Updated Response Assessment Criteria for High-Grade Gliomas: Response Assessment in Neuro-Oncology Work Group (RANO)
Time Frame: Up to 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Alisertib, Fractionated Stereotactic Radiosurgery
Number analyzed (Participants) | 17
Participants | 0

3. Secondary Outcome: Number of Participants With Progression Free Survival at 6 Months
Description: Estimated through the Kaplan-Meier method.
Time Frame: At 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Alisertib, Fractionated Stereotactic Radiosurgery
Number analyzed (Participants) | 17
Participants | 6

4. Secondary Outcome: Number of Participants With Overall Survival at 6 Months
Description: Estimated through the Kaplan-Meier method.
Time Frame: At 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Alisertib, Fractionated Stereotactic Radiosurgery
Number analyzed (Participants) | 17
Participants | 15

ADVERSE EVENTS:
Time Frame: 18 months from baseline
Arm/Group | Alisertib, Fractionated Stereotactic Radiosurgery
All-Cause Mortality (participants affected / at risk) | 15/17
Serious Adverse Events (participants affected / at risk) | 6/17
Other Adverse Events (participants affected / at risk) | 17/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Alisertib, Fractionated Stereotactic Radiosurgery (N=17)
Leukopenia (Blood and lymphatic system disorders) | 2
Neutropenia (Blood and lymphatic system disorders) | 2
Lymphopenia (Blood and lymphatic system disorders) | 1
Headache (Nervous system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Alisertib, Fractionated Stereotactic Radiosurgery (N=17)
Leukopenia (Blood and lymphatic system disorders) | 5
Neutropenia (Blood and lymphatic system disorders) | 1
Lymphopenia (Blood and lymphatic system disorders) | 7
Anemia (Blood and lymphatic system disorders) | 6
Transaminitis (Hepatobiliary disorders) | 2
Hyperlipidemia (Blood and lymphatic system disorders) | 4
Hyperbilirubinemia (Hepatobiliary disorders) | 3
Hyperglycemia (Metabolism and nutrition disorders) | 2
Hpocalcemia (Metabolism and nutrition disorders) | 5
Hyponatremia (Metabolism and nutrition disorders) | 2
Focal seizure (Nervous system disorders) | 2
Headache (Nervous system disorders) | 3
Fall (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 2
Gait Disturbance (Nervous system disorders) | 4
Peripheral Edema (General disorders) | 3
Muscle Weakness (Musculoskeletal and connective tissue disorders) | 4
Fatigue (General disorders) | 13
Hypertension (Cardiac disorders) | 3
Alopecia (General disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-13): https://cdn.clinicaltrials.gov/large-docs/09/NCT02186509/Prot_SAP_000.pdf